CLINICAL TRIAL: NCT05704166
Title: Pirfenidone Versus Placebo as Prophylaxis Against Acute Radiation-induced Lung Injury Following Hypofractionated Radiotherapy in Breast Cancer Patients (PRILI): A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study Evaluating
Brief Title: PirfenidoneVsPlacebo as Prophylaxis Against Acute Radiation-induced Lung Injury Following HFRT in Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Yang, Chief physician, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMUUH-BC-2201
Record Dates: First submitted 2022-12-21; First posted 2023-01-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Acute Lung Injury; Prevention
Keywords: Pirfenidone; Prophylaxis; Acute Radiation-induced Lung Injury; Breast Cancer
MeSH Terms: conditions — Acute Lung Injury; Breast Neoplasms | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The biostatistician (Chen Jinhua), who is not related to the statistical analysis of the data management performed in this experiment, used statistical software on the computer to generate random number tables by simple randomization according to the ratio of 1:1 between the experimental group and the control group. According to the existing random number table, the drug was coded by personnel unrelated to this study under the supervision of the clinical trial institution of the unit, and the random number and drug number assigned by the researcher according to the order of case enrollment were administered. The random number table and drug code are sealed together in the blind base as confidential data, and the blind base is kept in two sealed copies in the drug clinical research institution of the sponsor and the main investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pirfenidone (Experimental): Patients were given placebo or pirfenidone capsules orally one week before radiotherapy, 200mg/ time, 3 times a day in the first week; 300mg/ time 3 times daily for the second week and 400mg/ time 3 times daily for the third to eighth week. Take it after a meal.
  Interventions: Drug: Pirfenidone/Placebo
- Placebo (Placebo Comparator): Patients were given placebo or pirfenidone capsules orally one week before radiotherapy, 200mg/ time, 3 times a day in the first week; 300mg/ time 3 times daily for the second week and 400mg/ time 3 times daily for the third to eighth week. Take it after a meal.
  Interventions: Drug: Pirfenidone/Placebo

INTERVENTIONS:
Drug: Pirfenidone/Placebo — Patients were given drugs orally one week before radiotherapy, 200mg/ time, 3 times a day in the first week; 300mg/ time 3 times daily for the second week and 400mg/ time 3 times daily for the third to eighth week. Take it after a meal.
  Other Names: Pirfenidone Capsules/Placebo

SUMMARY:
The incidence of chest CT manifestations of lung injury after radiotherapy for breast cancer is more than 50%. Although the prognosis and quality of life of patients are rarely affected, it is still necessary to prevent the occurrence of minor radiation lung injury with the use of more novel drugs and subsequent salvage treatment may aggravate the radiation injury. This study intends to conduct a randomized, double-blind, single-center clinical study of pirfenidone versus placebo in the prevention of acute radiation induced lung injury after breast cancer surgery

DETAILED DESCRIPTION:
The incidence of chest CT manifestations of lung injury after radiotherapy for breast cancer is more than 50%. Although the prognosis and quality of life of patients are rarely affected, it is still necessary to prevent the occurrence of minor radiation lung injury with the use of more novel drugs and subsequent salvage treatment may aggravate the radiation injury. This study intends to conduct a randomized, double-blind, single-center clinical study of pirfenidone versus placebo in the prevention of acute radiation induced lung injury after breast cancer surgery.In this study, the incidence of grade 1-4 radiation lung injury was expected to be 60% in the radiotherapy alone group (placebo group), and pirfenidone capsules (experimental group) were expected to reduce the incidence of lung injury after radiotherapy to 40%. Bilateral test showed a statistical efficacy of 0.8 (α option 0.05). In this study, two independent rate comparison sample sizes were used to calculate, Binomial Enumeration method was used for 97 patients in both groups, and the expected shedding rate was 10%. 107 patients were needed in each group, and the total sample size was 214. Biological specimens are expected to be obtained from more than 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in this study, patients must meet all of the following inclusion criteria:

  1. Breast invasive carcinoma or ductal carcinoma in situ or lobular carcinoma in situ confirmed by histology;
  2. Age 18-75, female;
  3. The physical state score of the Eastern Tumor Cooperative Group (ECOG) was 0-2;
  4. Patients meeting the indications of postoperative radiotherapy and neoadjuvant chemotherapy: clinical stage 3 or above or postoperative ypT3-T4 or N+; Non-neoadjuvant chemotherapy patients: postoperative pathological staging of pT3-T4 or pN2 or above, or positive for upper and lower clavicle and lymph nodes in the internal milk region, or positive for clinical consideration; For patients with pT1-2N1, postoperative adjuvant radiotherapy should be determined based on the patient's age, tumor grade, incisal margin, number of positive lymph nodes, molecular typing, past complications, and patient's intention.
  5. Radiotherapy regimen was chest wall + supraclavicular 40Gy/15f after root modification, or whole milk ± upper and lower clavicular 40Gy/15f after breast preservation, tumor bed simultaneous supplement 50Gy/15f;
  6. All screening period laboratory tests should be performed in accordance with protocol requirements and within 28 days prior to enrollment. The values of laboratory tests performed by screening must meet the following criteria:

     blood routine check all meet the following criteria: A. Hb≥90g/L; B. ANC≥1.5×109/L; C. PLT≥70×109/L; biochemical examination all meet the following criteria: TBIL < 1.5× upper limit of normal range (ULN); ALT and AST≤2.5 x ULN; Serum Cr≤1.25×ULN or endogenous creatinine clearance ≥45 mL/min (Cockcroft-Gault formula)
  7. Women who are at risk of becoming pregnant must undergo a negative serum pregnancy test within 7 days before the first dose and be willing to use a highly effective method of contraception during the trial period and 120 days after the last dose of the test drug. Male subjects with a partner of a woman of reproductive age should be surgically sterilized or consent to a highly effective method of contraception during the trial period and 120 days after the last test drug administration;
  8. The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Patients with any of the following criteria were not enrolled in this study

  1. History and complications A. male breast cancer patients; B. Did not meet the conditions of large segmentation radiotherapy (upper and lower clavicular lymph node metastasis, internal milk lymph node metastasis, the patient refused large segmentation radiotherapy); C. The subject has any active, known, or suspected autoimmune disease. To admit subjects who are in a stable state and do not require systemic immunosuppressive therapy; D. The patient is participating in another clinical study or less than 4 weeks after the end of the previous clinical study; E. Patients with a known or highly suspected history of interstitial pneumonia; Or may interfere with the detection or management of suspected drug-related pulmonary toxicity; F. A history of other malignant tumors; Except in patients who have had potentially curable therapy and have not had disease recurrence for 5 years since treatment began; G. Pregnant women and patients with mental illness; H. Prior treatment with radiotherapy, chemotherapy, etc.; I. Patients with active tuberculosis should be excluded; J. Severe acute or chronic lung infections requiring systemic treatment; K. Patients with obvious blood coughing or daily hemoptysis of half a teaspoon (2.5ml) or more in the 2 months before randomization; L. Patients with heart failure (New York Heart Association standard Class III or IV), poor coronary artery disease control or arrhythmia, or a history of myocardial infarction in the 6 months prior to screening despite receiving appropriate medication.
  2. Physical examination and laboratory examination A. A known history of testing positive for human immunodeficiency virus (HIV) or a known history of acquired immunodeficiency syndrome (AIDS); B. untreated active hepatitis (hepatitis B: HBsAg positive with HBV DNA≥ 500 IU/mL; Hepatitis C: HCV RNA positive and abnormal liver function); Combined with hepatitis B and hepatitis C co-infection.
  3. As determined by the investigator, the patient may have other factors that may lead to the termination of the study, such as other serious diseases or serious abnormalities in laboratory tests or other factors that may affect the safety of the subjects, or family or social factors such as the collection of test data and samples.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female only
Enrollment: 214 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in lung injury grading on chest computerized tomography within 3 months after radiotherapy | 4 weeks and 12 weeks after radiotherapy
  Kouloulias scale was used to evaluate the changes of lung injury grading in chest computerized tomography within 3 months after radiotherapy. The higher the grading is, the more serious the lung injury is

SECONDARY OUTCOMES:
Relationship between biomarkers and radioactive damage | 1 week before medication，4 weeks and 12 weeks after radiotherapy
  The changes of the above cytokines in the blood of patients were monitored before and after radiotherapy, and the correlation between the changes of cytokines and the grade of radiation damage was analyzed
Relationship between biomarkers and therapy | 1 week before medication，4 weeks and 12 weeks after radiotherapy
  The changes of the above cytokines in the blood of patients were monitored before and after radiotherapy, and the correlation between the changes of cytokines and treatment was analyzed
security | Every week of the medication，4 weeks and 12 weeks after radiotherapy
  use the CTCAE5.0 scale to record adverse events to assess safety

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yang, Doctor, Principal Investigator — Director of the radiotherapy department
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Overgaard M, Jensen MB, Overgaard J, Hansen PS, Rose C, Andersson M, Kamby C, Kjaer M, Gadeberg CC, Rasmussen BB, Blichert-Toft M, Mouridsen HT. Postoperative radiotherapy in high-risk postmenopausal breast-cancer patients given adjuvant tamoxifen: Danish Breast Cancer Cooperative Group DBCG 82c randomised trial. Lancet. 1999 May 15;353(9165):1641-8. doi: 10.1016/S0140-6736(98)09201-0. PMID 10335782
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Overgaard M, Nielsen HM, Tramm T, Hojris I, Grantzau TL, Alsner J, Offersen BV, Overgaard J; DBCG Radiotherapy Group. Postmastectomy radiotherapy in high-risk breast cancer patients given adjuvant systemic therapy. A 30-year long-term report from the Danish breast cancer cooperative group DBCG 82bc trial. Radiother Oncol. 2022 May;170:4-13. doi: 10.1016/j.radonc.2022.03.008. Epub 2022 Mar 11. PMID 35288227
- [Background] Wang SL, Fang H, Hu C, Song YW, Wang WH, Jin J, Liu YP, Ren H, Liu J, Li GF, Du XH, Tang Y, Jing H, Ma YC, Huang Z, Chen B, Tang Y, Li N, Lu NN, Qi SN, Yang Y, Sun GY, Liu XF, Li YX. Hypofractionated Versus Conventional Fractionated Radiotherapy After Breast-Conserving Surgery in the Modern Treatment Era: A Multicenter, Randomized Controlled Trial From China. J Clin Oncol. 2020 Nov 1;38(31):3604-3614. doi: 10.1200/JCO.20.01024. Epub 2020 Aug 11. PMID 32780661
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Background] Offersen BV, Alsner J, Nielsen HM, Jakobsen EH, Nielsen MH, Krause M, Stenbygaard L, Mjaaland I, Schreiber A, Kasti UM, Overgaard J; Danish Breast Cancer Group Radiation Therapy Committee. Hypofractionated Versus Standard Fractionated Radiotherapy in Patients With Early Breast Cancer or Ductal Carcinoma In Situ in a Randomized Phase III Trial: The DBCG HYPO Trial. J Clin Oncol. 2020 Nov 1;38(31):3615-3625. doi: 10.1200/JCO.20.01363. Epub 2020 Sep 10. PMID 32910709
- [Background] Vicini FA, Cecchini RS, White JR, Arthur DW, Julian TB, Rabinovitch RA, Kuske RR, Ganz PA, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Costantino JP, Bear HD, Germain I, Gustafson G, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Bryant JL, Wolmark N. Long-term primary results of accelerated partial breast irradiation after breast-conserving surgery for early-stage breast cancer: a randomised, phase 3, equivalence trial. Lancet. 2019 Dec 14;394(10215):2155-2164. doi: 10.1016/S0140-6736(19)32514-0. Epub 2019 Dec 5. PMID 31813636
- [Background] Jung W, Shim SS, Kim K. CT findings of acute radiation-induced pneumonitis in breast cancer. Br J Radiol. 2021 Aug 1;94(1124):20200997. doi: 10.1259/bjr.20200997. Epub 2021 Jun 16. PMID 34111374
- [Background] Liu Y, Wang W, Shiue K, Yao H, Cerra-Franco A, Shapiro RH, Huang KC, Vile D, Langer M, Watson G, Bartlett G, Ai H, Sheski F, Jin JY, Zellars R, Fu P, Lautenschlaeger T, Kong FS. Risk factors for symptomatic radiation pneumonitis after stereotactic body radiation therapy (SBRT) in patients with non-small cell lung cancer. Radiother Oncol. 2021 Mar;156:231-238. doi: 10.1016/j.radonc.2020.10.015. Epub 2020 Oct 21. PMID 33096168
- [Background] Li F, Liu H, Wu H, Liang S, Xu Y. Risk factors for radiation pneumonitis in lung cancer patients with subclinical interstitial lung disease after thoracic radiation therapy. Radiat Oncol. 2021 Apr 13;16(1):70. doi: 10.1186/s13014-021-01798-2. PMID 33849579
- [Background] Jiang W, Song Y, Sun Z, Qiu J, Shi L. Dosimetric Factors and Radiomics Features Within Different Regions of Interest in Planning CT Images for Improving the Prediction of Radiation Pneumonitis. Int J Radiat Oncol Biol Phys. 2021 Jul 15;110(4):1161-1170. doi: 10.1016/j.ijrobp.2021.01.049. Epub 2021 Feb 3. PMID 33548340
- [Background] Hope AJ, Lindsay PE, El Naqa I, Alaly JR, Vicic M, Bradley JD, Deasy JO. Modeling radiation pneumonitis risk with clinical, dosimetric, and spatial parameters. Int J Radiat Oncol Biol Phys. 2006 May 1;65(1):112-24. doi: 10.1016/j.ijrobp.2005.11.046. PMID 16618575
- [Background] Mehta V. Radiation pneumonitis and pulmonary fibrosis in non-small-cell lung cancer: pulmonary function, prediction, and prevention. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):5-24. doi: 10.1016/j.ijrobp.2005.03.047. PMID 15963660
- [Background] Andreassen CN, Overgaard J, Alsner J, Overgaard M, Herskind C, Cesaretti JA, Atencio DP, Green S, Formenti SC, Stock RG, Rosenstein BS. ATM sequence variants and risk of radiation-induced subcutaneous fibrosis after postmastectomy radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):776-83. doi: 10.1016/j.ijrobp.2005.09.014. Epub 2005 Dec 9. PMID 16338099
- [Background] Tsoutsou PG, Koukourakis MI. Radiation pneumonitis and fibrosis: mechanisms underlying its pathogenesis and implications for future research. Int J Radiat Oncol Biol Phys. 2006 Dec 1;66(5):1281-93. doi: 10.1016/j.ijrobp.2006.08.058. PMID 17126203
- [Background] Puthawala K, Hadjiangelis N, Jacoby SC, Bayongan E, Zhao Z, Yang Z, Devitt ML, Horan GS, Weinreb PH, Lukashev ME, Violette SM, Grant KS, Colarossi C, Formenti SC, Munger JS. Inhibition of integrin alpha(v)beta6, an activator of latent transforming growth factor-beta, prevents radiation-induced lung fibrosis. Am J Respir Crit Care Med. 2008 Jan 1;177(1):82-90. doi: 10.1164/rccm.200706-806OC. Epub 2007 Oct 4. PMID 17916808
- [Background] Kim JY, Kim YS, Kim YK, Park HJ, Kim SJ, Kang JH, Wang YP, Jang HS, Lee SN, Yoon SC. The TGF-beta1 dynamics during radiation therapy and its correlation to symptomatic radiation pneumonitis in lung cancer patients. Radiat Oncol. 2009 Nov 27;4:59. doi: 10.1186/1748-717X-4-59. PMID 19943923
- [Background] Libshitz HI, Shuman LS. Radiation-induced pulmonary change: CT findings. J Comput Assist Tomogr. 1984 Feb;8(1):15-9. doi: 10.1097/00004728-198402000-00003. PMID 6690504
- [Background] Jenkins P, Welsh A. Computed tomography appearance of early radiation injury to the lung: correlation with clinical and dosimetric factors. Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):97-103. doi: 10.1016/j.ijrobp.2010.05.017. Epub 2011 May 3. PMID 21543163
- [Background] Kouloulias V, Zygogianni A, Efstathopoulos E, Victoria O, Christos A, Pantelis K, Koutoulidis V, Kouvaris J, Sandilos P, Varela M, Aytas I, Gouliamos A, Kelekis N. Suggestion for a new grading scale for radiation induced pneumonitis based on radiological findings of computerized tomography: correlation with clinical and radiotherapeutic parameters in lung cancer patients. Asian Pac J Cancer Prev. 2013;14(5):2717-22. doi: 10.7314/apjcp.2013.14.5.2717. PMID 23803021
- [Background] Kashihara T, Nakayama Y, Ito K, Kubo Y, Okuma K, Shima S, Nakamura S, Takahashi K, Inaba K, Murakami N, Igaki H, Ohe Y, Kusumoto M, Itami J. Usefulness of Simple Original Interstitial Lung Abnormality Scores for Predicting Radiation Pneumonitis Requiring Steroidal Treatment After Definitive Radiation Therapy for Patients With Locally Advanced Non-Small Cell Lung Cancer. Adv Radiat Oncol. 2020 Oct 31;6(1):100606. doi: 10.1016/j.adro.2020.10.019. eCollection 2021 Jan-Feb. PMID 33665489
- [Background] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Background] Yorke ED, Jackson A, Rosenzweig KE, Braban L, Leibel SA, Ling CC. Correlation of dosimetric factors and radiation pneumonitis for non-small-cell lung cancer patients in a recently completed dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Nov 1;63(3):672-82. doi: 10.1016/j.ijrobp.2005.03.026. Epub 2005 Jun 4. PMID 15939548
- [Background] Tsujino K, Hirota S, Kotani Y, Kado T, Yoden E, Fujii O, Soejima T, Adachi S, Takada Y. Radiation pneumonitis following concurrent accelerated hyperfractionated radiotherapy and chemotherapy for limited-stage small-cell lung cancer: Dose-volume histogram analysis and comparison with conventional chemoradiation. Int J Radiat Oncol Biol Phys. 2006 Mar 15;64(4):1100-5. doi: 10.1016/j.ijrobp.2005.09.025. Epub 2005 Dec 20. PMID 16373082
- [Background] Bradley JD, Hope A, El Naqa I, Apte A, Lindsay PE, Bosch W, Matthews J, Sause W, Graham MV, Deasy JO; RTOG. A nomogram to predict radiation pneumonitis, derived from a combined analysis of RTOG 9311 and institutional data. Int J Radiat Oncol Biol Phys. 2007 Nov 15;69(4):985-92. doi: 10.1016/j.ijrobp.2007.04.077. Epub 2007 Aug 6. PMID 17689035
- [Background] Shaverdian N, Shepherd AF, Rimner A, Wu AJ, Simone CB 2nd, Gelblum DY, Gomez DR. Need for Caution in the Diagnosis of Radiation Pneumonitis During the COVID-19 Pandemic. Adv Radiat Oncol. 2020 May 5;5(4):617-620. doi: 10.1016/j.adro.2020.04.015. eCollection 2020 Jul-Aug. PMID 32377597
- [Background] Wang YY, Tian XC, Zhu L, Bai XH, Zhao R. Concomitant Radiation Recall Dermatitis and Radiation Recall Pneumonitis Induced by Pembrolizumab. J Thorac Oncol. 2020 Oct;15(10):e160-e162. doi: 10.1016/j.jtho.2020.05.014. No abstract available. PMID 32981602
- [Background] Cousin F, Desir C, Ben Mustapha S, Mievis C, Coucke P, Hustinx R. Incidence, risk factors, and CT characteristics of radiation recall pneumonitis induced by immune checkpoint inhibitor in lung cancer. Radiother Oncol. 2021 Apr;157:47-55. doi: 10.1016/j.radonc.2021.01.001. Epub 2021 Jan 14. PMID 33453313
- [Background] De Giglio A, Scorsetti M, Franceschini D, Massari F, Ardizzoni A. Bilateral radiation recall pneumonitis during immunotherapy for an advanced renal cell carcinoma: A challenging case enhances the need for a multidisciplinary approach. Eur J Cancer. 2021 Jan;143:75-77. doi: 10.1016/j.ejca.2020.10.024. Epub 2020 Dec 7. No abstract available. PMID 33279856
- [Background] Noble PW, Albera C, Bradford WZ, Costabel U, Glassberg MK, Kardatzke D, King TE Jr, Lancaster L, Sahn SA, Szwarcberg J, Valeyre D, du Bois RM; CAPACITY Study Group. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet. 2011 May 21;377(9779):1760-9. doi: 10.1016/S0140-6736(11)60405-4. Epub 2011 May 13. PMID 21571362
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Neighbors M, Cabanski CR, Ramalingam TR, Sheng XR, Tew GW, Gu C, Jia G, Peng K, Ray JM, Ley B, Wolters PJ, Collard HR, Arron JR. Prognostic and predictive biomarkers for patients with idiopathic pulmonary fibrosis treated with pirfenidone: post-hoc assessment of the CAPACITY and ASCEND trials. Lancet Respir Med. 2018 Aug;6(8):615-626. doi: 10.1016/S2213-2600(18)30185-1. Epub 2018 Jun 29. PMID 30072107
- [Background] Behr J, Prasse A, Kreuter M, Johow J, Rabe KF, Bonella F, Bonnet R, Grohe C, Held M, Wilkens H, Hammerl P, Koschel D, Blaas S, Wirtz H, Ficker JH, Neumeister W, Schonfeld N, Claussen M, Kneidinger N, Frankenberger M, Hummler S, Kahn N, Tello S, Freise J, Welte T, Neuser P, Gunther A; RELIEF investigators. Pirfenidone in patients with progressive fibrotic interstitial lung diseases other than idiopathic pulmonary fibrosis (RELIEF): a double-blind, randomised, placebo-controlled, phase 2b trial. Lancet Respir Med. 2021 May;9(5):476-486. doi: 10.1016/S2213-2600(20)30554-3. Epub 2021 Mar 30. PMID 33798455
- [Background] Simone NL, Soule BP, Gerber L, Augustine E, Smith S, Altemus RM, Mitchell JB, Camphausen KA. Oral pirfenidone in patients with chronic fibrosis resulting from radiotherapy: a pilot study. Radiat Oncol. 2007 May 31;2:19. doi: 10.1186/1748-717X-2-19. PMID 17540023
- [Background] Sun YW, Zhang YY, Ke XJ, Wu XJ, Chen ZF, Chi P. Pirfenidone prevents radiation-induced intestinal fibrosis in rats by inhibiting fibroblast proliferation and differentiation and suppressing the TGF-beta1/Smad/CTGF signaling pathway. Eur J Pharmacol. 2018 Mar 5;822:199-206. doi: 10.1016/j.ejphar.2018.01.027. Epub 2018 Jan 31. PMID 29374548
- [Background] Qin W, Liu B, Yi M, Li L, Tang Y, Wu B, Yuan X. Antifibrotic Agent Pirfenidone Protects against Development of Radiation-Induced Pulmonary Fibrosis in a Murine Model. Radiat Res. 2018 Oct;190(4):396-403. doi: 10.1667/RR15017.1. Epub 2018 Jul 17. PMID 30016220